CLINICAL TRIAL: NCT00173667
Title: A Randomized Controlled Study of Nifecardia SRFC (Nifedipine) and Adalat OROS (Nifedipine) in the Treatment of Patients With Essential Hypertension
Brief Title: A Study of Nifecardia SRFC and Adalat OROS in the Treatment of Patients With Essential Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 182CL1
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nifedipine

INTERVENTIONS:
Drug: Nifedipine 30 mg GITS

SUMMARY:
Objective:

* To evaluate the antihypertensive efficacy of two brands of nifedipine 30mg in patients with hypertension.
* To assess the safety of 8 weeks of therapy with two brands of nifedipine 30mg in patients with hypertension.
* To study flow-mediated dilatation and oxidative stress in nonsmoker with essential hypertension but without diabetes mellitus or dyslipidemia.

Study Design:

* Head-to-head, randomized and parallel design.
* A total of 60 patients with a clinically confirmed diagnosis of hypertension will provide 30 available patients in each treatment group.
* The drugs and dosage will be as follows:

Group A: nifedipine 30-60mg once daily (Nifecardia, CCPC) Group B: nifedipine 30-60 mg once daily (Adalat OROS, Bayer)

Method:

After washout period, the eligible patients will randomly be allocated to receive two brands of nifedipine 30 mg once daily. Each patient will receive two times of ambulatory blood pressure measurement (ABPM) at both entrance and final stages of the study. The patients will also undergo complete clinical evaluation. Therapy dosage will be started at a dose of nifedipine 30 mg once daily. Dosage will be adjusted if systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg by office measurement after 4 weeks of treatment. Nifedipine will be increased to 60 mg once daily. The Ambulatory blood pressure measurement will be set to take reading at 1-hour intervals during the 24 hours assessment.

Physical examination included the measurement of heart rate and blood pressure. The value will be read on Visit 1 and 3-12 hours after the last dose of nifedipine. Routine laboratory test includes hematology, blood chemistry and urinalysis. Hematology test and fasting blood chemistry test will be measured immediately before the start of treatment and after 8 weeks' treatment or at time of discontinuation. Thiobarbituric acid-reactive substances (TBARS) in patient plasma were measured for oxidative stress and endothelium-dependent flow-mediated vasodilation will also be evaluated. Possible concomitant medication will remain constant throughout the study. The physician will question the patients as to their compliance at each visit. If compliance dose not reach 80%, the subject will be dropped out.

DETAILED DESCRIPTION:
1. Introduction:

Nifedipine is one of the first calcium-channel blockers that are widely used in the treatment of hypertension. Because of its long-term application experience and safety profile, traditional nifedipine has been remodeled as a sustained released formulary of Nifecardia SRFC. Nifecardia SRFC is a new formulary designed of zero-order kinetic release system that maintain a constant plasma concentration of nifedipine and achieve the target of once daily application. Nifecardia SRFC is bioequivalence in efficacy with that of Adalat OROS which is also a sustained released type of calcium-channel blockers. In this study, the efficacy and safety profile of Nifecardia SRFC and Adalat OROS will be evaluated with randomized head-to-head design to treat the patients with hypertension.

2. Objective:

1. To evaluate the antihypertensive efficacy of two brands of nifedipine (30mg) in patients with hypertension.
2. To assess the safety of 8 weeks of therapy with two brands of nifedipine (30mg) in patients with hypertension.
3. To study flow-mediated dilatation and oxidative stress in nonsmoker with essential hypertension but without diabetes mellitus or dyslipidemia.

3. Study Design:

1. Head-to-head, randomized and parallel design.
2. A total of 60 patients with a clinically confirmed diagnosis of hypertension will provide 30 available patients in each treatment group.

   Inclusion criteria are:
   * Male or non-pregnant female patients aged 18-70 years.
   * Patients had hypertension with sitting systolic blood pressure 140-180 mmHg, or diastolic blood pressure 90-110 mmHg.
   * Patients must give written informed consent to participate in this study.

   Exclusion criteria are:
   * Women who are pregnant or nursing.
   * Patients have the evidence of secondary or malignant hypertension, history of severe heart disease, cerebrovascular accident within one year, or myocardial infarction within six months.
   * Patients receiving more than one anti-hypertensive agents or one antihypertensive agent with maximal recommended dosage before entrance into the trial.
   * Patients with uncontrolled diabetes mellitus.
   * Patients had known hypersensitivity or contraindication to nifedipine, other calcium channel blockers or other beta-adrenergic antagonists.
   * Patients have the evidences of hepatic dysfunction (AST, ALT> 3 times upper limit of normal value), renal dysfunction (serum creatinine concentration>1.5 mg/dl), pulmonary dysfunction, mental disorders or other concurrent severe disease.
   * As to the study of flow-mediated dilatation and oxidative stress, patients with diabetes mellitus, dyslipidemia, body mass index >27, and smokers will be excluded.
3. The drugs and dosage will be as follows:

Group A: nifedipine 30-60mg once daily (Nifecardia, CCPC) Group B: nifedipine 30-60 mg once daily (Adalat OROS, Bayer)

4. Method:

After washout period, the eligible patients will randomly be allocated to receive two brands of nifedipine 30 mg once daily. Each patient will receive two times of ambulatory blood pressure measurement (ABPM) at both entrance and final stages of the study. The patients will also undergo complete clinical evaluation. Therapy dosage will be started at a dose of nifedipine 30 mg once daily. Dosage will be adjusted if systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg by office measurement after 4 weeks of treatment. Nifedipine will be increased to 60 mg once daily. The Ambulatory blood pressure measurement will be set to take reading at 1-hour intervals during the 24 hours assessment.

Physical examination included the measurement of heart rate and blood pressure. The value will be read on Visit 1 and 3-12 hours after the last dose of nifedipine. Routine laboratory test includes hematology, blood chemistry and urinalysis. Hematology test and fasting blood chemistry test will be measured immediately before the start of treatment and after 8 weeks' treatment or at time of discontinuation. Thiobarbituric acid-reactive substances (TBARS) in patient plasma were measured for oxidative stress and endothelium-dependent flow-mediated vasodilation will also be evaluated. Possible concomitant medication will remain constant throughout the study. The physician will question the patients as to their compliance at each visit. If compliance dose not reach 80%, the subject will be dropped out.

Withdrawal of a subject is based on the following three assessments: (1) not compliant with study protocol, (2) occurrence of severe symptoms or complications, (3) unacceptable side effects with the study drug.

5. Adverse event and Safety evaluation:

All adverse events will be recorded in the adverse event section of case report form (CRF). Serious drug adverse events will be notified within 24h to hospital and the monitor of China Chemistry& Pharmaceuticals Co. Safety evaluation is based on doctor's evaluation on the results of clinical laboratory test and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female patients aged 18-70 years.
* Patients had hypertension with sitting systolic blood pressure 140-180 mmHg, or diastolic blood pressure 90-110 mmHg.
* Patients must give written informed consent to participate in this study.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Patients have the evidence of secondary or malignant hypertension, history of severe heart disease, cerebrovascular accident within one year, or myocardial infarction within six months.
* Patients receiving more than one anti-hypertensive agents or one antihypertensive agent with maximal recommended dosage before entrance into the trial.
* Patients with uncontrolled diabetes mellitus.
* Patients had known hypersensitivity or contraindication to nifedipine, other calcium channel blockers or other beta-adrenergic antagonists.
* Patients have the evidences of hepatic dysfunction (AST, ALT> 3 times upper limit of normal value), renal dysfunction (serum creatinine concentration>1.5 mg/dl), pulmonary dysfunction, mental disorders or other concurrent severe disease.
* As to the study of flow-mediated dilatation and oxidative stress, patients with diabetes mellitus, dyslipidemia, body mass index >27, and smokers will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Overall Officials: Gen-Gae Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Cardiovascular Division, Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan